CLINICAL TRIAL: NCT07087002
Title: Phase I Clinical Trial of GPC2 Chimeric Antigen Receptor T (GPC2-CAR T) Cells for Relapsed or Refractory Medulloblastoma in Children and Young Adults
Brief Title: GPC2-CAR T Cell Therapy for Relapsed or Refractory Medulloblastoma in Children and Young Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-79066; NCI-2025-06836 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2025-06-24; First posted 2025-07-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Medulloblastoma; Central Nervous System Embryonal Tumor; Refractory Medulloblastoma; Recurrent Medulloblastoma; Pediatric Brain Tumor; Embryonal Tumor With Multilayered Rosettes (ETMR); Pineoblastoma; Atypical Teratoid/Rhabdoid Tumor (ATRT) of the CNS; CNS Neuroblastoma; FOXR2-activated
Keywords: GPC2-CAR T cells; Chimeric Antigen Receptor T cells; Intracerebroventricular CAR T; Pediatric CNS tumors; Immunotherapy; Medulloblastoma; Refractory brain tumors; T cell therapy; Embryonal Tumor with Multilayered Rosettes (ETMR); Pineoblastoma; Atypical Teratoid/Rhabdoid Tumor (ATRT) of the CNS; CNS neuroblastoma; FOXR2-activated
MeSH Terms: conditions — Medulloblastoma; Neuroectodermal Tumors, Primitive; Pinealoma; Rhabdoid Tumor; Brain Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GPC2-CAR T Cell Therapy (Experimental): Participants will undergo leukapheresis for collection of peripheral blood mononuclear cells, which will be used to manufacture autologous T cells transduced with a retroviral vector encoding a GPC2-targeted chimeric antigen receptor (GPC2-CAR T cells). After lymphodepleting chemotherapy with fludarabine and cyclophosphamide, participants will receive up to 8 cycles of intracerebroventricular (ICV) GPC2-CAR T cell infusions using an intrapatient dose escalation strategy.
  Interventions: Biological: GPC2-CAR T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: GPC2-CAR T cells — Autologous T cells transduced with retroviral vector encoding a second-generation GPC2-targeted chimeric antigen receptor (GPC2-CAR), administered intracerebroventricularly. Up to 8 doses are given every 28 days, following an intrapatient dose escalation schema.
  Other Names: GPC2-directed CAR T cells
Drug: Fludarabine — Administered as part of a lymphodepleting chemotherapy regimen prior to GPC2-CAR T cell infusion. Dose: 30 mg/m²/day for 3 days.
Drug: Cyclophosphamide — Administered with fludarabine for lymphodepletion. Dose: 500 mg/m²/day for 3 days.

SUMMARY:
This is a single-site, open-label Phase 1 clinical trial evaluating the feasibility, safety, and preliminary activity of autologous GPC2-targeted chimeric antigen receptor (CAR) T cells administered via intracerebroventricular (ICV) infusion in children and young adults with relapsed or refractory medulloblastoma or other eligible Central Nervous System (CNS) embryonal tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Histologically confirmed diagnosis of medulloblastoma or other primary CNS embryonal tumor according to 2021 CNS WHO Classification (5th edition)

   * Other acceptable CNS embryonal tumors include:
   * Embryonal Tumor with Multilayered Rosettes (ETMR)
   * Pineoblastoma
   * Atypical Teratoid/Rhabdoid Tumor (ATRT) of the CNS
   * CNS neuroblastoma, FOXR2-activated
   * CNS Embryonal Tumor NOS
2. Recurrent/Refractory Disease: History of relapsed and/or recurrent disease defined as tumor progression or recurrence following initial diagnosis and upfront treatment with curative intent, or failure to achieve disease control with standard curative-intent therapy.
3. GPC2 Positive: H-score ≥ 100 by IHC staining performed on the (Prescreening Protocol IRB-78780, PI: Katherine Ryan, DO) at Stanford Clinical Anatomic Pathology Lab for GPC2 from a tumor sample any time since initial diagnosis.
4. Evaluable Disease: Evaluable disease as per radiographic findings and/or positive cerebrospinal fluid cytology within 28 days of enrollment.
5. Patients with VP shunts: Patients with pre-existing ventriculo-peritoneal (VP) shunt devices must have a programmable shunt device to enroll on this study. A VP shunt is not a requirement for this study.
6. Prior therapy: No limit to the number of prior treatment regimens. Toxicities due to prior therapy must be stable or recovered to ≤ Grade 1 (except for clinically non-significant toxicities such as alopecia, nutritional support measures, electrolyte abnormalities, or those not impacting the investigator's ability to assess treatment emergent toxicities).

   At time of enrollment, subjects are on track to meet the required therapy wash out period(s) prior to apheresis.

   a. At least 6 weeks following craniospinal radiation therapy. i. At least 14 days wash-out needed following small volume radiotherapy (i.e., Stereotactic Radiosurgery (SRS)).

   b. At least 21 days or 5 half-lives (whichever is shorter) must have elapsed since any prior systemic therapy, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half-lives.

   c. At least 28 days following bevacizumab treatment. d. At least 30 days following any investigational drug. e. At least 12 weeks following systemic inhibitory or stimulatory immune checkpoint therapy.
7. Age: ≥ 12 months to ≤ 30 years of age at time of enrollment The first 3 subjects treated with GPC2-CAR T cells must be ≥ 3 years old at time of infusion
8. Performance Status: Subjects ≥ 16 years of age must have Karnofsky ≥ 60%. Subjects < 16 years of age must have Lansky scale 60%; or ECOG performance status ≤ 2 (see Section 11.3).
9. Normal Organ and Marrow Function [supportive care is allowed per institutional standards, i.e., filgrastim, transfusion]

   1. Hemoglobin ≥ 8 g/dL
   2. Absolute Neutrophil Count (ANC) ≥ 1,000/μL
   3. Platelet count ≥ 75,000/μL, with no platelet transfusion within 96 hours prior to enrollment
   4. Absolute lymphocyte count (ALC) ≥ 150/μL
   5. PT/INR, PTT ≤ 1.5 x ULN for age

      Adequate renal, hepatic, cardiac, and pulmonary function defined as:
   6. Serum creatinine < 1.5 x ULN for age and gender, OR creatinine clearance or GFR (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m2
   7. Serum ALT or AST ≤ 3x ULN
   8. Total bilirubin ≤ 1.5 mg/dL, unless subject has Gilbert's Syndrome
   9. Cardiac ejection fraction ≥ 45%
   10. No evidence of physiologically significant pericardial effusion as determined by an ECHO
   11. No clinically significant ECG findings
   12. No clinically significant pleural effusion
   13. Pulse oximetry ≥ 92% on room air, OR forced vital capacity ≥ 50% of predicted value
10. Not Pregnant: Females of childbearing potential must have a negative pregnancy test.
11. Contraception: Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) months after receiving the preparative regimen or for as long as CAR T cells are detectable in peripheral blood.
12. Must provide informed consent. All subjects ≥ 18 years of age must be able to give informed consent. For subjects <18 years old or adults with limited decision-making capacity, their legal authorized representative (LAR) (i.e., parent or guardian) must give informed consent. Pediatric subjects will be included in age-appropriate discussion and assent will be obtained for those > 7 years of age, when appropriate. If a minor becomes of age during participation of this study, he/she will be asked to reconsent as an adult.

Exclusion Criteria

1. Any patient with metastatic disease OUTSIDE the CNS.
2. Unwilling or unable, in the investigator's judgement, to have a CSF reservoir (Ommaya or Rickham) placed. Does not apply to subjects who have a pre-existing device suitable for ICV delivery of CAR T cells and ICP monitoring.
3. Clinical evidence of active/on-going significant increased intracranial pressure (i.e., impending herniation) or uncontrolled seizures.
4. Prior receipt of a chimeric antigen receptor (CAR)-based therapy.
5. Currently receiving anticoagulation therapy.
6. Known history of infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive).

   EXCEPTION: A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
7. Pregnancy or breastfeeding in a postpartum female.
8. Known sensitivity or allergy to any agents/reagents used in this study.
9. History of prior other malignancy. EXCEPTION: Previously diagnosed and definitively treated more than 5 years prior to enrollment or whose prognosis is deemed good enough to not warrant surveillance.
10. Primary immunodeficiency or history of autoimmune disease (e.g., Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
11. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
12. Significant medical diseases or poorly controlled conditions that, in the judgement of the investigator, put the subject at an unacceptable risk of complications, including but not limited to: uncontrolled diabetes mellitus, chronic obstructive pulmonary disease, pulmonary fibrosis, clinically significant inflammatory disorders, immunodeficiency (e.g., HIV infection), immunocompromised for reasons other than malignancy (e.g., chronic corticosteroid therapy or other immunosuppressive therapy), renal failure including patients requiring dialysis, or clinically significant liver dysfunction.
13. In the Investigator's judgment, the subject or parents/caregivers (as required) will not be able to comply with the study procedures outlined in the study protocol including follow-up visits.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Manufacturing Feasibility | Up to 6 months post-leukapheresis
  Proportion of manufacturing attempts that result in at least one dose of GPC2-CAR T cells that meet the IND release criteria and protocol-specified dose.
Incidence of Dose Limiting Toxicities (DLTs) | Within first 28-day treatment cycle per dose level
  Number and severity of DLTs following GPC2-CAR T cell administration at each dose level using protocol-defined criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years post-infusion
  Percentage of subjects achieving a protocol-defined response (complete response, partial response, or stable disease) based on imaging and neurological exam.
Progression-Free Survival (PFS) | Up to 2 years
  Time from enrollment to radiographic disease progression.
Overall Survival (OS) | Up to 2 years
  Time from initial diagnosis to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ryan, DO, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States